CLINICAL TRIAL: NCT06465030
Title: Identification of Pattern and Factors Affecting Recurrence of Head and Neck Carcinoma After Radical IMRT and VMAT
Brief Title: Identification of Pattern and Factors Affecting Recurrence in Head and Neck Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reem Gamal Mohamed, RESIDENT, Sohag University
Other Study IDs: Soh-Med-24-04-017MS
Record Dates: First submitted 2024-05-29; First posted 2024-06-18 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The study will evaluate the local experiences in treatment of head and neck carcinoma by retrospectively analyzing the incidence and location of recurrence, and also studying factors affecting this recurrence.

DETAILED DESCRIPTION:
The investigators will evaluate the local experience in treatment of head and neck SCC by retrospectively analyzing the incidence and location of recurrence, either; local recurrence (LR), regional recurrence (RR), or distant mets in eligible head and neck cancer patients treated with IMRT and VMAT in the period from 2018 till 2022 to allow a follow-up for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged more than 18 years. Patients with primary non nasopharyngeal head and neck squamous cell carcinoma. Patients who were intended to receive radical treatment delivered by IMRT and VMAT techniques.

Exclusion Criteria:

* Adults who had double malignancies. Metastatic HNSCC cases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent head and neck cancer after radical treatment by IMRT and VMAT, in Sohag city.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pattern of relapse in recurrent head and neck squamous cell carcinoma, evident clinically and measured by images "US,CT, MRI and endoscopy". | At least obsevation of 1 year FU of the patient
  Local, locoregional recurrence by MRI neck and CT Neck and distant recurrence by pan CTs.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Gamal, M.B.B.Ch, Principal Investigator — Sohag university hospital, oncology and nuclear medicine department
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt